CLINICAL TRIAL: NCT03755128
Title: A Multicenter, Prospective Observational Study to Characterize the Clinical Course of Pregnant Women and Children at High Risk for Early Onset Severe Hemolytic Disease of the Fetus and Newborn
Brief Title: A Study to Characterize the Clinical Course of Pregnant Women and Children at High Risk for Early Onset Severe Hemolytic Disease of the Fetus and Newborn
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR109067; MOM-M281-103 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-11-26; First posted 2018-11-27 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Early Onset Severe Hemolytic Disease of the Fetus and Newborn (EOS-HDFN); Erythroblastosis, Fetal
Keywords: Hemolytic disease of the fetus and newborn (HDFN); Erythroblastosis, Fetal; Early onset severe hemolytic disease of the fetus and newborn (EOS-HDFN); M281; Pregnant Women
MeSH Terms: conditions — Erythroblastosis, Fetal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women and their offspring from current pregnancy
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No investigational drugs will be administered as part of the study

SUMMARY:
The primary purpose of the study is to characterize the current standard of care, clinical course, and outcomes of pregnant women and their offspring at high risk for early onset severe hemolytic disease of the fetus and newborn (EOS-HDFN).

DETAILED DESCRIPTION:
The outcomes of interest will be assessed from the information collected on the standard of care treatment for EOS-HDFN in pregnant women and their offspring from current pregnancy.

ELIGIBILITY:
Pregnant female participants must be ≥18 years of age with an estimated Gestational Age of ≥ 8 weeks; not currently pregnant with multiples (twins or more); and no other clinically relevant abnormalities currently or in their history that the Investigator would deem them ineligible to participate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants must have an obstetrical history of severe fetal anemia, hydrops, or stillbirth related to hemolytic disease of the fetus and newborn, have alloantibody titers for anti-D ≥32 or anti-Kell titers ≥4, and be currently pregnant with an antigen-positive fetus. Eligible women may enter the study at any time during the current pregnancy prior to delivery.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Live Birth at or After Gestational Age (GA) Week 32 Without Intrauterine Transfusion (IUT) | GA Week 32 through GA Week 37

SECONDARY OUTCOMES:
Percentage of Participants With Live Birth | Up to approximately GA Week 37
Percentage of Participants at GA Week 24 Without an IUT | Week 24
GA at First IUT | Up to approximately GA Week 37
Number of IUTs Required | Up to approximately GA Week 37
Percentage of Participants With Fetal Hydrops | Post-Birth through Age 3 Months
Percentage of Neonates Requiring Phototherapy | Post-Birth through Age 3 Months
Percentage of Neonates Requiring Exchange Transfusions | Post-Birth through Age 3 Months
Number of days of phototherapy required by neonate | Post-Birth through Age 3 Months
Percentage of Neonates Requiring Simple Transfusions in the First 3 Months of Life | Post-Birth through Age 3 Months
Number of Simple Transfusions Required by Neonate in the First 3 Months of Life | Post-Birth through Age 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (18):
- United States (5):
  - Columbia University Medical Center, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - UPMC, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- Australia (2):
  - Liverpool Hospital, Liverpool
  - The Royal Women's Hospital, Parkville
- Universitair Ziekenhuis Leuven, Leuven, Belgium
- Canada (3):
  - The University of British Columbia, Vancouver, British Columbia
  - Mount Sinai Hospital, Toronto, Ontario
  - Centre Hospitalier Sainte Justine, Montreal, Quebec
- Justus-Liebig-Universität Gießen, Kinderherzzentrum, Giessen, Germany
- Leiden University Medical Center, Leiden, Netherlands
- Spain (2):
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Univ. San Cecilio, Granada
- Karolinska Universitetssjukhuset Huddinge, Stockholm, Sweden
- United Kingdom (2):
  - Queen Elizabeth Hospital, Edgbaston
  - University College London Hospitals NHSFT, London